CLINICAL TRIAL: NCT02570113
Title: A Post-Market Study of Transcatheter Perivascular Renal Denervation for the Treatment of Hypertension Using the Ablative Solutions Inc. Peregrine System™ Infusion Catheter
Brief Title: The Peregrine Post-Market Study for the Treatment of Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ablative Solutions, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR0001
Record Dates: First submitted 2015-10-06; First posted 2015-10-07 (Estimated); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renal Denervation by Neurolysis (Experimental): Infusion of 0.6 ml of dehydrated alcohol (not less than 95% by volume) into the peri-adventitial space of the renal artery, to achieve renal denervation by neurolysis, via three simultaneous deployed needles, situated at the distal end of the Peregrine System Infusion Catheter.
  Interventions: Device: Peregrine System Infusion Catheter

INTERVENTIONS:
Device: Peregrine System Infusion Catheter — The Peregrine Catheter is inserted bilaterally into the renal arteries and a specified amount of a neurolytic agent is inserted into the vessel walls.

SUMMARY:
The Ablative Solutions, Inc. Peregrine System Infusion Catheter is a catheter-based device which is intended to be used to ablate the afferent and efferent sympathetic nerves serving the kidneys. The catheter is inserted via the femoral artery, steered into the renal artery, and then delivers, by infusion from its distal end, a neurolytic agent. This targets the nerve bundles, which are in the adventitia - a sheath surrounding the artery. The aim is to reduce blood pressure in cases of hypertension, including seriously elevated blood pressure which does not respond to drug treatment. This study will evaluate the safety and performance of the device.

DETAILED DESCRIPTION:
There is strong evidence in the published literature that the renal nerves are important contributors to hypertension, and that their ablation does not have adverse side-effects.

The literature provides technical, clinical and scientific evidence supporting the use of perivascular renal denervation for a carefully defined patient group.

An existing device (the Medtronic Symplicity catheter) was initially shown to be safe and effective for achieving perivascular renal denervation by delivery of radio-frequency energy. The results of early nonrandomized clinical studies (HTN-1, HTN-2) found that perivascular renal denervation by radio-frequency energy delivery was an effective therapy, associated with very low risks. In other contexts, denervation can also be safely and effectively achieved by neurolytic agents.

The ASI Peregrine System™ Infusion Catheter and the denervation procedure in general is similar enough to the Medtronic Symplicity catheter to enable the use of published data to establish the validity of the design concept of the Peregrine System and estimate the likely levels of risk of side effects. It can be concluded from the literature that the ASI Peregrine System™ will achieve percutaneous renal denervation with a low risk of procedural complications (comparable to accepted percutaneous interventional therapies) and without long-term impairment of renal artery or kidney function or other serious adverse events.

Previous premarket clinical trials have provided support for the safe and effective use of the Peregrine Catheter for the treatment of patients with hypertension. The Peregrine System Infusion Catheter is currently CE marked and the indication for use is "The Peregrine System™ Infusion Catheter is intended for the infusion of a neurolytic agent to achieve a reduction in systemic blood pressure in hypertensive patients." Based upon the literature and previous clinical data, chemical denervation is an appropriate treatment for the specified study population of adults who have hypertension despite taking at least 3 anti-hypertensive drugs of different classes including at least one diuretic.

The objectives of this post-market study are to collect additional safety and performance data pertaining to renal denervation by using dehydrated alcohol as a chemical neurolytic agent delivered into the adventitial/peri-adventitial area of the renal arteries for the purpose of renal denervation, using the Peregrine System™ Infusion Catheter, in patients with hypertension.

In order for the study to be valid, only one chemical neurolytic agent can be used. The Coordinating Investigator has chosen to use dehydrated alcohol (not less than 95% by volume) for therapeutic neurolysis, therefore all participating sites will use this agent.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subject, age 18-80, male or female;
2. Subject has a target treatment vasculature diameter of ≥4 mm and ≤ 7 mm and length of ≥5 mm;
3. Subject has 3 measurements with a mean of office Systolic Blood Pressure of

   ≥150 mmHg AND office Diastolic Blood Pressure of ≥85 mmHg;
4. Subject has a 24-hour mean systolic Ambulatory Blood Pressure Measurement (ABPM) ≥135 mm Hg with ≥70% valid readings (as determined by measurement device);
5. Subject with hypertension is receiving and adhering to a stable medication regimen of at least 3 anti-hypertensive medications of different classes (for at least 4 consecutive weeks), one of which must be a diuretic;
6. Subject agrees to have all study procedures performed, to comply with medication regimen and is able and willing to comply with all study follow-up visits;
7. Subject has provided written informed consent.

Exclusion Criteria:

1. Subject has a contraindication known for conventional percutaneous interventional procedures such as:

   * intolerance for antiplatelet/anticoagulant therapy
   * known allergy to contrast media
   * bleeding disorders (such as bleeding diathesis, thrombocytopenia and severe anemia)
2. Subject has documented severe untreated obstructive sleep apnea (Apnea Hypopnea Index [AHI] ≥30 per hour);
3. Subjects with nephrotic syndrome;
4. Subjects on immunosuppressive medications or immunosuppressive doses of steroids;
5. Subject has type 1 diabetes mellitus;
6. Subject is pregnant or nursing or planning to become pregnant;
7. Subject has an eGFR ≤20 mL/min/1.73m2

   , based on the CKD-EPI equation;
8. Subject has imaging-assessed renal artery anatomy abnormalities or variations based on Investigator's evaluation of the screening images [i.e. MRA/CTA examination and/or renal angiography]) meeting one of the following criteria:

   * Renal artery stenosis >60% of the normal diameter segment (diameter stenosis, compared to the angiographically normal proximal or distal segment);
   * Any renal artery abnormality or disease that, per the physician assessment, precludes the safe insertion of the guiding catheter (such as but not limited to severe renal artery aneurysm, excessive tortuosity, severe renal artery calcification);
   * Previous renal angioplasty associated with stenting or other implants, that, per the physician's assessment, precludes the safe deployment of the Peregrine catheter components in the target treatment segment of the renal artery;
9. Subject has a history of nephrectomy, a single kidney or kidney tumor, or urinary tract obstruction (with potential for hydronephrosis);
10. Subject is known to have a non-functioning kidney or unequal renal size (>2 cm difference in renal length between kidneys associated with a chronic kidney disease or a deterioration of the kidney function);
11. Subject has a renal transplant;
12. Subject has a history of myocardial infarction, unstable angina pectoris, or stroke/TIA within the last six months from planned procedure;
13. Subject has hemodynamically significant valvular heart disease;
14. Subject has heart failure (NYHA III or IV) or has an ejection fraction ≤30%;
15. Subject with chronic atrial fibrillation;
16. Subjects who are allergic or intolerant of the neurolytic agent (such as dehydrated alcohol);
17. Any contraindication to the imaging as required per the protocol;
18. Subject has a life expectancy of <12 months;
19. Subject is currently enrolled in other potentially confounding research, i.e., another therapeutic or interventional research trial. Subjects enrolled in observational registries may still be eligible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-11; Primary Completion 2019-02 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Horst Sievert, MD, Principal Investigator — CardioVasculares Centrum (CVC) Frankfurt
Locations (10):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- Na Homolce Hospital, Prague, Czechia
- Germany (6):
  - Charite-Universitaetsmedizin Berlin, Berlin
  - Universitätsklinik Erlangen Klinik für Nephrologie/Hypertensiologie, Erlangen
  - Elisabeth-Krankenhause, Essen
  - CardioVasculares Centrum (CVC) Frankfurt, Frankfurt
  - Universitats-Herzzentrum/University Heart Center Klinik fur Kardiologie und Angiologie, Freiburg im Breisgau
  - Klinik fur Innere Medizin III, Homburg
- Poland (2):
  - Oddzial Kardiologii Inwazyjnej, Tychy
  - Oddizal Kardiologiczno-Angiologiczny PAKS, Ustroń

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mahfoud F, Sievert H, Bertog S, Lauder L, Ewen S, Lengele JP, Wojakowski W, Schmieder R, van der Giet M, Weber MA, Kandzari DE, Parise H, Fischell TA, Pathak A, Persu A. Long-Term Results up to 12 Months After Catheter-Based Alcohol-Mediated Renal Denervation for Treatment of Resistant Hypertension. Circ Cardiovasc Interv. 2021 Sep;14(9):e010075. doi: 10.1161/CIRCINTERVENTIONS.120.010075. Epub 2021 Sep 2. PMID 34470501

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Withdrawal of consent (N=3)
Period: Overall Study
Arm/Group | Renal Denervation by Neurolysis
Started | 45
Completed | 42
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Renal Denervation by Neurolysis
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Europe | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With the Absence of Particular Events as Adjudicated by the CEC Through 1-month Post Procedure:
Description: The primary safety endpoint is defined by the absence of any of the following events as adjudicated by the CEC through 1-month post procedure:
  1. Peri-procedural major vascular complications;
  2. Major Bleeding as defined by the TIMI Bleeding Classification;
  3. Acute Kidney Injury (AKI) within 1 month of the procedure
  4. Peri-procedural death (within 1 month of the procedure)
Time Frame: 1-month
Measure: Number; unit: participants
Arm/Group | Renal Denervation by Neurolysis
Number analyzed (Participants) | 45
participants | 43

2. Primary Outcome: Change in 24-hour Mean Ambulatory Systolic Blood Pressure From Baseline to 6 Months
Description: The primary performance endpoint is defined as a reduction of 24-hour mean ambulatory systolic blood pressure following treatment at 6 months, as compared to baseline.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation by Neurolysis
Number analyzed (Participants) | 42
mmHg | -11 (14)

3. Secondary Outcome: Numbr of Subjects With a Decline in eGFR by >25% From Baseline to 6 Months
Description: Proportion of subjects with a decline in eGFR by >25% from baseline to 6-month follow-up;
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation by Neurolysis
Number analyzed (Participants) | 44
Participants | 2

4. Secondary Outcome: Change in Serum Creatinine From Baseline to 6 Months
Description: Change in serum creatinine from baseline to 6-month follow-up
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Renal Denervation by Neurolysis
Number analyzed (Participants) | 44
mg/dL | 0.01 (0.13)

5. Secondary Outcome: Number of Participants With New Renal Arterial Stenosis > 60%
Description: Number of Participants with New renal arterial stenosis > 60% from the baseline at the 6-month follow-up, to be confirmed by the same imaging method used at baseline.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation by Neurolysis
Number analyzed (Participants) | 44
Participants | 0

6. Secondary Outcome: Number of Subjects With Stroke or Transient Ischemic Attack (TIA) With 1 Month of the Procedure
Description: Stroke or TIA within 1 month of the procedure
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation by Neurolysis
Number analyzed (Participants) | 45
Participants | 0

7. Secondary Outcome: Number of Subjects With Myocardial Infarction (MI) Within 1 Month of the Procedure
Description: Myocardial Infarction (MI) within 1 month of the procedure
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation by Neurolysis
Number analyzed (Participants) | 45
Participants | 0

8. Secondary Outcome: Number of Participants With Major Adverse Events (MAE) Through 6 Months Post-Procedure
Description: Number of Participants with Major Adverse Events (MAE) through 6-month post-procedure. MAE is defined as the occurrence of any of the following:
  1. All-cause death
  2. End stage renal failure
  3. Significant embolic event resulting in end-organ damage or requiring intervention to prevent it
  4. Major Vascular Complications (including major artery dissections)
  5. Significant new renal artery stenosis (>60% diameter stenosis)
  6. Hypertensive crisis (hypertensive emergency only)
  7. Severe hypotension/syncope
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation by Neurolysis
Number analyzed (Participants) | 44
Participants | 3

9. Secondary Outcome: Changes in Antihypertensive Medications at 7 Days, and 1, 3, 6 and 12 Months Post-Procedure
Description: Changes in antihypertensive medications at 7-day, 1, 3, 6 and 12 months post procedure;
Time Frame: 7-day, 1, 3, 6 and 12 months
Reporting Status: Not Posted

10. Secondary Outcome: Changes in Systolic and Diastolic Clinic/Office Blood Pressure
Description: Changes in systolic and diastolic clinic/office blood pressure following treatment compared to baseline, assessed at 7-day, 1, 3, 6 and 12 months post-procedure.
Time Frame: 7-day, 1, 3, 6 and 12 months
Reporting Status: Not Posted

11. Secondary Outcome: Changes in Systolic and Diastolic 24-hour Mean Daytime and Nighttime Ambulatory Blood Pressure
Description: Changes in systolic and diastolic 24-hour mean daytime and nighttime ambulatory blood pressure, assessed at 1, 3, 6 and 12-month post-procedure.
Time Frame: 1, 3, 6 and 12-months
Reporting Status: Not Posted

12. Secondary Outcome: Changes in Diastolic 24-hour Mean Ambulatory Blood Pressure
Description: Changes in systolic and diastolic 24-hour mean ambulatory blood pressure assessed at 1, 3, 6 and 12-month post-procedure.
Time Frame: 1, 3, 6 and 12-months
Reporting Status: Not Posted

13. Secondary Outcome: Changes in Systolic 24-hour Mean Ambulatory Blood Pressure
Description: Changes in systolic 24-hour mean ambulatory blood pressure assessed at 1, 3 and 12 months postprocedure;
Time Frame: 1, 3 and 12 months
Reporting Status: Not Posted

14. Secondary Outcome: Change in eGFR
Description: Change in eGFR from baseline, to evaluate the progression of Chronic Kidney Disease (CKD) after 1, 3, 6 and 12 months;
Time Frame: 1, 3, 6 and 12 months
Reporting Status: Not Posted

15. Secondary Outcome: The Progression of Kidney Disease
Description: The progression of kidney disease in subjects with ≤60 mL/min/1.73m2 will be evaluated by comparing the change in eGFR during the study to the historical loss (reduction) of eGFR during the 3 years prior to renal denervation for each individual subject;
Time Frame: 1, 3, 6, and 12 months
Reporting Status: Not Posted

16. Secondary Outcome: Change in Albuminuria
Description: Change in albuminuria from baseline to 3 months post-procedure, with additional assessments at each study time point;
Time Frame: 3, 6, and 12 months
Reporting Status: Not Posted

17. Secondary Outcome: Change in Albuminuria Categorization
Description: Change in albuminuria categorization from baseline to 3 months post-procedure, with additional assessments at each study time point;
Time Frame: 3, 6, and 12 months
Reporting Status: Not Posted

18. Secondary Outcome: Change in Serum Creatinine and Cystatin-C
Description: Change in serum creatinine and cystatin-C from baseline to 3 months postprocedure, with additional assessments at each study time point.
Time Frame: 3, 6, and 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Renal Denervation by Neurolysis
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 11/45
Other Adverse Events (participants affected / at risk) | 42/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Denervation by Neurolysis (N=45)
haematoma (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Vascular access site infection (Infections and infestations) | 1 (1)
Psychiatric evaluation (Investigations) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Ureteral stent removal (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Renal Denervation by Neurolysis (N=45)
hematoma (Vascular disorders) | 12
back pain (Musculoskeletal and connective tissue disorders) | 11
vertigo (Ear and labyrinth disorders) | 5
upper respiratory tract infection (Infections and infestations) | 4
headache (Nervous system disorders) | 4
bradycardia (Cardiac disorders) | 4
nausea (Gastrointestinal disorders) | 3
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
arrhythmia (Cardiac disorders) | 3
nasopharyngitis (Infections and infestations) | 3
vascular pseudoaneurysm (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/13/NCT02570113/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT02570113/SAP_001.pdf